CLINICAL TRIAL: NCT01403779
Title: Comparison of the Cosmetic Outcome of Hypofractionated Versus Normofractionated Intensity Modulated Radiotherapy (IMRT) in Treatment of Breast Cancer: The KOSIMA Trial
Brief Title: Comparison of the Cosmetic Outcome of Hypofractionated Versus Normofractionated IMRT in Treatment of Breast Cancer
Acronym: KOSIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Prof. Dr., Universitätsmedizin Mannheim
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-KOSIMA-01; ARO 2010-3 (Other: Arbeitsgemeinschaft Radiologische Onkologie der Deutschen Krebsgesellschaft)
Record Dates: First submitted 2010-10-29; First posted 2011-07-27 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Tumors; Breast Cancer
Keywords: Intensity-Modulated Radiation Therapy (IMRT); Breast cancer; Hypofractionation
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Hypofractionated IMRT (Active Comparator): hypofractionated IMRT for right sided breast cancer
  Interventions: Radiation: intensity modulated radiotherapy (IMRT) for breast cancer
- 2-Normofractioated IMRT (Active Comparator): normofractionated IMRT for left sided breast cancer
  Interventions: Radiation: intensity modulated radiotherapy (IMRT) for breast cancer

INTERVENTIONS:
Radiation: intensity modulated radiotherapy (IMRT) for breast cancer — right sided breast cancer patients are stratified to receive a hypofractionated treatment course (40.05 / 2.67Gy in 15 fractions) and the left sided breast cancer patients a normofractionated irradiation (50/2Gy in 25 fractions). In both arms, patients between 60-69 years are to receive a boost (16 Gy / 2Gy).
  Other Names: Arm 1, Arm 2

SUMMARY:
Several multicenter studies have shown the equivalence of hypofractionated radiotherapy and normofractionated radiotherapy after breast-conserving surgery. However, the treatment in these studies was carried out with conventional techniques and not with the modern IMRT. Also the evaluation of quality of life and cosmetic outcome were not standardized.

This study is a two-arm prospective study comparing normofractionated and hypofractionated radiotherapy in patients with breast cancer using tangential IMRT techniques.

The primary endpoints are acute and chronic cosmetic breast changes. The secondary endpoint is the patients' quality of life.

Patients to be included are breast cancer 60 years old patients or older with tumour stages pTis-pT3, pN0-pN1a, M0 after breast-conserving surgery. Patients with right sided breast cancer are stratified to receive a hypofractionated treatment course (40.05 / 2.67Gy in 15 fractions) and the left sided breast cancer a normofractionated irradiation (50/2Gy in 25 fractions). In both arms, patients between 60-69 years are to receive a boost (16 Gy / 2Gy).

In both groups, a tangential intensity-modulated radiation technique aiming to achieve optimal dose homogeneity is applied.

Since higher single radiation dose to the heart can lead to higher morbidity and/or mortality, patient stratification according to the diseased side was adopted where the left-sided breast cancer patients would receive normofractionated 2Gy single dose. Therefore there is no randomization.

For classification and grading of adverse cosmetic events, the "Common Toxicity Criteria (CTC-AE V3.0) and the recognized LENT-SOMA scores are to be regularly documented. Quality of life is to be documented with two standardized, validated questionnaires "QLQ C30 and BR23" of the EORTC (European Organization for Research and Treatment of Cancer). The questionnaires are to be filled by the patients themselves at different time points during the study period.

A sum of grade III fibrosis, grade III telangiectasia and grade II hyperpigmentation of around 20% is expected after 2 years.

Therefore, calculation of the required number of cases based on an alpha of 0.05 and a power of 80% with a maximal tolerable toxicity difference of 15% within 2 years results in the need for recruiting 226 patients (113 in each arm) (non-inferiority of hypofractionated therapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive or in situ breast cancer, tumor stage pTis-pT3, pN0-1a, M0
* Age ≥ 60 years
* signed informed consent from the patient

Exclusion Criteria:

* Stage pN1b-PN3, pT4 and / or M1
* incomplete surgical resection
* after mastectomy of the ipsilateral or contralateral breast
* breast reconstruction with implant or expander insert
* bilateral breast cancer
* Lack of compliance or consent
* Indications for irradiation of the axillary, supraclavicular or parasternal lymph nodes

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2010-07; Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
acute and chronic cosmetic outcome | 2 years

SECONDARY OUTCOMES:
acute and chronic cosmetic outcome, Quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Wenz, MD, Study Chair — UMM
Locations (1):
- Department of Radiotherapy University Hospital Mannheim, Mannheim, Germany

REFERENCES:
- [Result] Sarria GR, Welzel G, Polednik M, Wenz F, Abo-Madyan Y. Prospective Comparison of Hypofractionated Versus Normofractionated Intensity-Modulated Radiotherapy in Breast Cancer: Late Toxicity Results of the Non-Inferiority KOSIMA Trial (ARO2010-3). Front Oncol. 2022 May 5;12:824891. doi: 10.3389/fonc.2022.824891. eCollection 2022. PMID 35600361
- See also: German Abstract — https://doi.org/10.1055/s-0033-1347536
- See also: English Abstract — http://dx.doi.org/10.1016/j.ijrobp.2013.06.552